CLINICAL TRIAL: NCT06663423
Title: Cohort Study on the Differential Impact of Anxiety and Depression on Implicit and Explicit Memory Performance
Brief Title: Impact of Anxiety and Depression on Implicit and Explicit Memory Performance
Acronym: ADEM
Status: Completed | Type: Observational
Sponsor: Islamic Azad University, Sanandaj (Other)
Responsible Party: Principal Investigator, Shaghayegh Radmehr, Principal Investigator, Department of Psychiatry, Tehran Institute of Psychiatry, Islamic Azad University, Sanandaj
Other Study IDs: SDU-MEMORY-2024
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Major Depressive Disorder (MDD); Generalized Anxiety Disorder (GAD); Memory Bias; Implicit Memory; Explicit Memory
Keywords: Anxiety; Depression; Cognitive Bias; Memory Processing; Emotional Influence on Memory; Word Recognition Task; Mood-Congruent Memory; Psychological Disorders
MeSH Terms: conditions — Depressive Disorder, Major; Generalized Anxiety Disorder; Anxiety Disorders; Depression; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1: Depressive Disorder group - 9 participants.
- Group 2: Generalized Anxiety Disorder group - 9 participants.
- Group 3: Control group - 9 participants.

SUMMARY:
This study examines the effect of anxiety and depression on memory processes, focusing on implicit and explicit memory. Implicit memory involves unconscious recall, such as recognizing familiar words without effort, while explicit memory requires conscious recollection of specific information. The study aims to investigate whether individuals with depression and anxiety show differences in these types of memory, which may contribute to biases related to their emotional states.

Participants were divided into three groups: individuals with depressive disorder, individuals with generalized anxiety disorder, and a control group with no emotional disorders. Each group was assessed using tasks designed to measure both implicit and explicit memory performance. The goal is to enhance understanding of memory biases in individuals with depression and anxiety, potentially supporting more targeted interventions.

DETAILED DESCRIPTION:
This cohort study is designed to explore potential memory biases in individuals with depressive and anxiety disorders compared to a control group. The study includes 27 participants divided into three groups: nine individuals diagnosed with major depressive disorder, nine with generalized anxiety disorder, and nine control subjects with no history of emotional disorders. All participants were matched by age and education level.

Participants completed standardized tasks and assessments, including the Spielberger State-Trait Anxiety Inventory and various memory tasks such as word decoding and recognition memory tasks. These tasks aim to evaluate mood-congruent biases in memory recall. Data collection will focus on analyzing any distinct memory processing patterns in depression and anxiety to improve psychological treatment approaches.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Individuals diagnosed with major depressive disorder (Group 1)
* Individuals diagnosed with generalized anxiety disorder (Group 2)
* Healthy individuals with no history of emotional disorders (Group 3)

Exclusion Criteria:

* History of neurological disorders
* Visual impairments
* Substance abuse or drug addiction
* Psychiatric hospitalizations unrelated to primary diagnosis (for Groups 1 and 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A sample of individuals from Tehran Institute of Psychiatry and Shahid Esmaili Clinic, including patients with depressive disorder, generalized anxiety disorder, and a control group of healthy individuals with no history of emotional disorders.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2024-08-10 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Explicit Memory Bias | At a single time point during the experimental session, approximately 1 day
  The primary outcome is to assess explicit memory bias by measuring word recognition in participants with depressive disorder, generalized anxiety disorder, and a control group. Word recognition accuracy and response times are evaluated to determine mood-congruent biases specific to each group.

SECONDARY OUTCOMES:
Implicit Memory Bias | At a single time point during the experimental session, approximately 1 hour
  Secondary outcome is to assess implicit memory bias using a tachistoscopic word recognition task, measuring participants' ability to identify emotionally congruent words (e.g., words associated with depression, anxiety, and neutral words) without conscious awareness.

OTHER OUTCOMES:
Mood Congruence in Recognition Performance | At a single time point during the experimental session, approximately 1 hour
  Analysis of mood-congruent recognition performance across different emotional word types (depression-related, anxiety-related, pleasant, and neutral) to determine if participants show selective attention based on mood.

CONTACTS AND LOCATIONS:
Locations (1):
- Tehran Institute of Psychiatry and/or Shahid Esmaili Clinic., Tehran, Tehran Province, Iran